CLINICAL TRIAL: NCT00438711
Title: Surgical Decision Making Among People With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI K07 CA104701; GCO#03-0141 (Other: Mt Sinai); K07CA104701 (NIH)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2011-07

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study for people with inflammatory bowel disease ("IBD"--that is, ulcerative colitis, Crohn's colitis, or indeterminate colitis). We are studying how people with IBD decide to have surgery when a doctor has told them they should think about having their colon (large bowel) removed. This surgery is called a "colectomy." Patients will be asked to fill out a questionnaire that takes about 60 to 90 minutes to complete. Questions ask about patients' background (age, etc.) and their IBD. They also ask about patients' decision to have surgery or not to have surgery. For instance, what kinds of things did they think about? Some questions ask about other people who affected the choice and how patients felt about the help they got from others. People who wish to join the study will receive payment to thank them for their time.

* Patients must be at least 18 years old
* Patients must speak English
* Patients must have been told by their doctor to think about having surgery to take out their colon to (a) lower their risk for cancer or (b) because they have pre-cancer (called "dysplasia")
* Patients do not need to have had the surgery--they may have already had the surgery, they may not have had it yet, or they may have decided they do not want to have it

ELIGIBILITY:
Inclusion Criteria:

1. Have been told by a doctor that they have ulcerative colitis, Crohn's disease, or indeterminate colitis.
2. Be at least 18 years old
3. Speak English
4. Have been told by a doctor to think about having surgery to take out their colon ("colectomy") within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with inflammatory bowel disease who respond to advertisements and study announcements or who were treatment at the recruitment site and referred by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rini, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States